CLINICAL TRIAL: NCT03428932
Title: Glycemic Control and the Brain in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Washington University School of Medicine (Other); Stanford University (Other); University of Iowa (Other); Yale University (Other); Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000766
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2019-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin pump; Closed loop; Brain development; Pediatric; Type 1 Diabetes; MRI; Cognitive development
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Care (Active Comparator): Subjects will continue on their current treatment (insulin pump or injections), with follow up every 3 months. Neurocognitive testing and brain MRI/fMRI will be done at enrollment and 6 months.
  Interventions: Other: Standard Care
- Closed-Loop (Active Comparator): Subjects will transition from their current treatment (insulin pump or injections) onto the Medtronic 670G insulin pump (intervention arm as a comparator) and will have close contact with the study team. Neurocognitive testing and brain MRI/fMRI will be done at enrollment and 6 months.
  Interventions: Device: Closed Loop (Medtronic 670G)

INTERVENTIONS:
Device: Closed Loop (Medtronic 670G) — A loaner Medtronic 670G insulin pump, Enlite 3 sensor and GST3C Guardian transmitter will be utilized
  Arms: Closed-Loop
Other: Standard Care — Subjects will continue on their current treatment (insulin pump or injections), with follow up every 3 months.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to determine if improving diabetes control by better controlling blood sugars, will help improve or normalize brain function as compared to routine diabetes care. We will use either the patient's own insulin routine (injections or insulin pumps) or a closed-loop insulin pump (Medtronic 670G). This system uses a continuous glucose monitor (CGM) and an insulin pump to automatically give insulin and may improve control of blood sugars.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 14 and not yet 18 years old
* Must have been diagnosed with T1D prior to 5 years old but after 6 months
* For those diagnosed prior to 1 year of age, a positive blood test for an antibody marker will be required
* Have been born term or near term (≥34 weeks) and weighed more than≥ 2 kg (4.4lbs) at birth
* Be in puberty

Exclusion Criteria:

* History of intellectual disability, language or learning disability identified before diagnosis of diabetes, or enrollment in a self-contained special education program
* ADD/ADHD and/or on stimulant medication
* Any known genetic or medical problem that could impair brain development
* Abnormalities of the brain/nervous system, visual or hearing problem
* History of seizures not associated with fever before diabetes diagnosis
* Previous inpatient psychiatric treatment
* Unable to have a MRI of the head due to having metal: including metal ear tubes, full set of braces in mouth (retainer is acceptable), other appliances, or vascular clip

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Nemours Childrens Clinic, Jacksonville, Florida
  - University of Iowa, Iowa City, Iowa
  - Washington University St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database will be placed in the public domain after the completion of the study. This will be timed if possible with publication of the manuscripts that will result from these studies. In addition, formal requests for data will be accepted and reviewed by the DirecNet Steering Committee. If the request is approved, the Data Coordinating Centers will provide the data in a format mutually agreeable to the requesting party.
Time Frame: After completion of the study

REFERENCES:
- [Background] Bjorgaas MR. Cerebral effects of severe hypoglycemia in young people with type 1 diabetes. Pediatr Diabetes. 2012 Feb;13(1):100-7. doi: 10.1111/j.1399-5448.2011.00803.x. Epub 2011 Jul 25. No abstract available. PMID 21790920
- [Background] Saggar M, Tsalikian E, Mauras N, Mazaika P, White NH, Weinzimer S, Buckingham B, Hershey T, Reiss AL; Diabetes Research in Children Network (DirecNet). Compensatory Hyperconnectivity in Developing Brains of Young Children With Type 1 Diabetes. Diabetes. 2017 Mar;66(3):754-762. doi: 10.2337/db16-0414. Epub 2016 Oct 4. PMID 27702833
- [Background] Hosseini SM, Mazaika P, Mauras N, Buckingham B, Weinzimer SA, Tsalikian E, White NH, Reiss AL; Diabetes Research in Children Network (DirecNet). Altered Integration of Structural Covariance Networks in Young Children With Type 1 Diabetes. Hum Brain Mapp. 2016 Nov;37(11):4034-4046. doi: 10.1002/hbm.23293. PMID 27339089
- [Background] Mazaika PK, Weinzimer SA, Mauras N, Buckingham B, White NH, Tsalikian E, Hershey T, Cato A, Aye T, Fox L, Wilson DM, Tansey MJ, Tamborlane W, Peng D, Raman M, Marzelli M, Reiss AL; Diabetes Research in Children Network (DirecNet). Variations in Brain Volume and Growth in Young Children With Type 1 Diabetes. Diabetes. 2016 Feb;65(2):476-85. doi: 10.2337/db15-1242. Epub 2015 Oct 28. PMID 26512024
- [Background] Mauras N, Mazaika P, Buckingham B, Weinzimer S, White NH, Tsalikian E, Hershey T, Cato A, Cheng P, Kollman C, Beck RW, Ruedy K, Aye T, Fox L, Arbelaez AM, Wilson D, Tansey M, Tamborlane W, Peng D, Marzelli M, Winer KK, Reiss AL; Diabetes Research in Children Network (DirecNet). Longitudinal assessment of neuroanatomical and cognitive differences in young children with type 1 diabetes: association with hyperglycemia. Diabetes. 2015 May;64(5):1770-9. doi: 10.2337/db14-1445. Epub 2014 Dec 8. PMID 25488901
- [Background] Cato MA, Mauras N, Ambrosino J, Bondurant A, Conrad AL, Kollman C, Cheng P, Beck RW, Ruedy KJ, Aye T, Reiss AL, White NH, Hershey T; Diabetes Research in Children Network (DirecNet). Cognitive functioning in young children with type 1 diabetes. J Int Neuropsychol Soc. 2014 Feb;20(2):238-47. doi: 10.1017/S1355617713001434. PMID 24512675
- [Background] Barnea-Goraly N, Raman M, Mazaika P, Marzelli M, Hershey T, Weinzimer SA, Aye T, Buckingham B, Mauras N, White NH, Fox LA, Tansey M, Beck RW, Ruedy KJ, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). Alterations in white matter structure in young children with type 1 diabetes. Diabetes Care. 2014 Feb;37(2):332-40. doi: 10.2337/dc13-1388. Epub 2013 Dec 6. PMID 24319123
- [Background] Perantie DC, Koller JM, Weaver PM, Lugar HM, Black KJ, White NH, Hershey T. Prospectively determined impact of type 1 diabetes on brain volume during development. Diabetes. 2011 Nov;60(11):3006-14. doi: 10.2337/db11-0589. Epub 2011 Sep 27. PMID 21953611
- [Background] Ly TT, Breton MD, Keith-Hynes P, De Salvo D, Clinton P, Benassi K, Mize B, Chernavvsky D, Place J, Wilson DM, Kovatchev BP, Buckingham BA. Overnight glucose control with an automated, unified safety system in children and adolescents with type 1 diabetes at diabetes camp. Diabetes Care. 2014 Aug;37(8):2310-6. doi: 10.2337/dc14-0147. Epub 2014 May 30. PMID 24879841
- [Background] Hovorka R, Elleri D, Thabit H, Allen JM, Leelarathna L, El-Khairi R, Kumareswaran K, Caldwell K, Calhoun P, Kollman C, Murphy HR, Acerini CL, Wilinska ME, Nodale M, Dunger DB. Overnight closed-loop insulin delivery in young people with type 1 diabetes: a free-living, randomized clinical trial. Diabetes Care. 2014;37(5):1204-11. doi: 10.2337/dc13-2644. PMID 24757227
- [Background] Gazdzinski S, Durazzo TC, Mon A, Yeh PH, Meyerhoff DJ. Cerebral white matter recovery in abstinent alcoholics--a multimodality magnetic resonance study. Brain. 2010 Apr;133(Pt 4):1043-53. doi: 10.1093/brain/awp343. Epub 2010 Feb 4. PMID 20133395
- [Derived] Reiss AL, Jo B, Arbelaez AM, Tsalikian E, Buckingham B, Weinzimer SA, Fox LA, Cato A, White NH, Tansey M, Aye T, Tamborlane W, Englert K, Lum J, Mazaika P, Foland-Ross L, Marzelli M, Mauras N; Diabetes Research in Children Network (DirecNet) Consortium. A Pilot randomized trial to examine effects of a hybrid closed-loop insulin delivery system on neurodevelopmental and cognitive outcomes in adolescents with type 1 diabetes. Nat Commun. 2022 Aug 30;13(1):4940. doi: 10.1038/s41467-022-32289-x. PMID 36042217

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two enrolled participants did not meet inclusion/exclusion criteria and were screen failures before randomization. Two additional participants failed to complete all required baseline assessments or procedures. The remaining 42 subjects participated in the study and were included in all data analyses in line with the intention to treat principle. There were no additional participant losses.
Period: Overall Study
Arm/Group | Standard Care | Closed-Loop
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Closed-Loop | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 21 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (0.97) | 15.9 (1.76) | 15.8 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 15 | 34
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42
Gray Matter Volume [Number; unit: cm^3] | 739.16 | 727.27 | 734.22

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gray Matter Volume in the Brain
Description: Trends in total and regional grey matter volume
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: centimeters cubed
Arm/Group | Standard Care | Closed-Loop
Number analyzed (Participants) | 21 | 21
centimeters cubed | -4.83 [-8.92 to -0.74] | -9.31 [-14.46 to -4.17]

2. Secondary Outcome: Changes in Brain Activation (Dorsal Anterior Cingulate, Inferior Frontal Gyrus and/or Parietal Cortex)
Description: Blood Oxygen level diffusion (BOLD) Functional Magnetic Resonance Imaging (fMRI) was measured to assess functional activation occurring during "no-go" relative to "go" trials during a Go/No-Go cognitive task. Parameter estimates for an individual subject are obtained by modeling the subject's BOLD time series at each voxel against the expected BOLD response to a given task. Statistical weights (i.e., parameter estimates of activation strength) are determined based on how closely the observed and expected signals agree for each task condition to create parameter maps over the entire brain. Higher-level parameter estimates are generated via contrasts of the estimates from specific task conditions, which can lead to positive or negative values, depending on the relative activation of the conditions.
Time Frame: 6 months
Population: fMRI was not available for 3 Subjects in the Standard Care Group and for 1 in the Closed-Loop Group.
Measure: Median (95% Confidence Interval); unit: parameter estimates (betas)
Arm/Group | Standard Care | Closed-Loop
Number analyzed (Participants) | 18 | 20
parameter estimates (betas) | 78.58 [35.98 to 158.81] | -119.51 [-297.01 to -104.65]

3. Secondary Outcome: Changes in WASI-II Perceptual Reasoning Index (PRI)
Description: The Wechsler Abbreviated Scale of Intelligence second edition (WASI-II) was used. The WASI-II is composed of four subtests: Block Design, Vocabulary, Matrix Reasoning, and Similarities. The WASI-II used in this study produces a Perceptual Reasoning Index (PRI) score from the Block Design and Matrix Reasoning subtests' age-corrected scaled scores. The index scores are derived from a summation of the comprising scaled scores. The PRI score range is: 50-150. Higher scores mean better outcomes. Change over time in the PRI score is reported in each group.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard Care | Closed-Loop
Number analyzed (Participants) | 21 | 21
score on a scale | 2.05 [-0.17 to 4.27] | 6.10 [4.05 to 8.14]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Care | Closed-Loop
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=21) | Closed-Loop (N=21)
Hyperglycemia, Large Ketones, DKA (Endocrine disorders) | 0 (0) | 1 (1)
Acute illness: Tonsillitis (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03428932/Prot_SAP_000.pdf